CLINICAL TRIAL: NCT00210392
Title: Phase II Study of VELCADE in Patients With Extranodal Marginal Zone B-Cell Lymphoma of MALT-Type Pretreated With More Than One Prior Systemic Therapy Regimen (X05142)
Brief Title: VELCADE in MALT Lymphoma Pretreated With More Than One Prior Systemic Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After IELSG25A study amendment, patients subject of the present study were eligible for inclusion in the IELSG25A study
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: International Extranodal Lymphoma Study Group (IELSG), IELSG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG25B
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma, Mucosa-Associated Lymphoid Tissue
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bortezomib (drug) — Bortezomib 1,3 mg/m2 iv d1,4,8,11 every 21 days. Total 6 cycles

SUMMARY:
The primary objective of this study is to assess the antitumor activity (in terms of overall response rate - ORR - i.e. sum of complete and partial responses) of bortezomib in pretreated MALT lymphomas with more than one prior systemic therapy regimen

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven diagnosis of marginal zone B-cell lymphoma of MALT type arisen at any extranodal site
2. any stage (Ann Arbor I-IV)
3. relapsed or refractory disease pretreated with > 1 prior chemotherapy regimen and/or anti-CD20 immunotherapy
4. no evidence of histologic transformation to a high grade lymphoma
5. measurable or evaluable disease
6. age > 18 years
7. full recovery from previous therapy, with life expectancy of at least 6 months
8. ECOG performance status 0-2
9. for primary gastric localized H. pylori-positive disease at diagnosis:

   1. persistent disease 1 year after documented H. pylori infection eradication
   2. clinical, endoscopic (or histologic) evidence of progression at any time after H. pylori infection eradication
10. no prior chemotherapy, immunotherapy or radiotherapy in the last 6 weeks
11. no corticosteroids during the last 4 weeks, unless prednisone chronically administered at a dose <20 mg/day for indications other than lymphoma or lymphoma-related symptoms
12. adequate renal function (calculated or measured creatinine clearance >30 mL/minute), liver function (ASAT/ALAT <2,5 upper normal, total bilirubin <2,5x upper normal) and bone marrow function
13. no evidence of active opportunistic infections
14. no known HIV infection
15. no active HBV and/or HCV infection
16. no serious medical illness likely to interfere with participation in this clinical study
17. voluntary written informed consent before performance of any study-related procedure
18. female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

1. prior diagnosis of neoplasm within 5 years, except cervical intraepithelial neoplasia type 1. (CIN1) or localized non-melanomatous skin cancer
2. other investigational drugs with 14 days before enrollment
3. evidence of symptomatic central nervous system (CNS) disease
4. severe impairment of bone marrow function (ANC <1.0x109/L, PLT <30x109/L within 14 days before enrollment), unless due to lymphoma involvement
5. evidence of ≥ grade 2 peripheral neuropathy within 14 days before enrollment
6. known hypersensitivity to bortezomib, boron or mannitol
7. pregnant or lactating status, confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women
8. any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Antitumor activity, in terms of overall response rate (ORR) i.e. sum of complete and partial responses | During treatment and one month after treatment completion

SECONDARY OUTCOMES:
Safety, as acute and long-term toxicity | 18 months after treatment completion
Response duration (RD) (time to relapse or progression) in responders | 18 months after treatment completion
Progression-free survival (PFS) (time to disease progression or death from lymphoma) in all patients | 18 months after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Franco Cavalli, Study Chair — International Extranodal Lymphoma Study Group
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland

REFERENCES:
- See also: Click here for more information about this study — http://www.ielsg.org